CLINICAL TRIAL: NCT05045924
Title: A Pilot Study of Remote Home Monitoring in Patients With Advanced Cirrhosis, During COVID-19, Using Wearable Technology and an App Based Interface, to Diagnose Early and Severe Cirrhosis Decompensation, and Inform Design of a Future Randomized Controlled Intervention Study.
Brief Title: CirrhoCare in COVID-19: A Pilot, Remote, Home Monitoring Study in Advanced Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: CirrhoCare
Record Dates: First submitted 2021-09-14; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: 20 patients with decompensated liver cirrhosis monitored using a wrist-watch wearable device, with associated smart weighing scales and blood pressure cuff, along with a smartphone application (including economic smartphone in those patients if not available), to facilitate home monitoring.
- Control group: 20 patients with decompensated liver cirrhosis receiving standard quality of care.

SUMMARY:
The COVID-19 outbreak has exposed many strengths and weaknesses of delivering healthcare, and we want to assess whether patients with advanced liver cirrhosis can be effectively monitored at home, to limit hospital visits and thereby their infection risks. We also wish to show that if they have new signs of clinical deterioration, that these can be picked up quickly even in the community, and can result in early review or appropriate treatment. This study has been funded by INNOVATE UK, who are seeking novel ways and technologies to improve health during the pressures of the COVID pandemic.

Taking part in this study involves a consultation with the investigating doctor and being shown how to use a phone-based App and the supplied CirrhoCare equipment (Withings Watch, scales, and Blood Pressure cuff). Patients will be shown how to use the equipment for several simple daily assessments, including:

Heart rate (ECG) readings via the supplied Withings Watch. This would take approximately 7-10 minutes to perform each day.

Daily weight, using a special weighing scale that also measures the amount of body water and muscle percentages (takes 30 seconds to perform).

Digital blood pressure measurement, using the supplied cuff. This would take approximately 2 minutes to perform daily.

For all the above measurements, that are entirely automated, the patient will be guided via the mobile phone App with step-by-step video instructions. In addition, they will be given printed instructions. Individuals will be asked to perform the measurements through daily prompts built into the App, and be sent reminders, in case they forget. If they have difficulties with any of the tasks, there is also an App based support system, where they can send a message for the trial team to provide assistance.

In addition to the measurements above, patients will be prompted to click on a memory testing exercise of naming animals (termed - 'Stroop test'), which will be performed after the daily morning measurements. This can take half a minute to up to four minutes to perform, depending on an individual's memory function.

The equipment will be supplied will enable daily monitoring for a maximum of 3 months in this study. We will also be able to learn from the supplied watch, how much sleep and how much daily exercise patients get, which will help us assess general physical well-being. Furthermore, patients will be aksed to supply information on the amount of fluid and food they have consumed via simple 'click' functions on the App (e.g. clicking next to the picture denoting 4 glasses of water). Patients will be prompted to do this via smartphone and watch every evening.

We will seek patient feedback on using the App through a brief in-App based questionnaire, after 4, 8 and 12 weeks of study. In addition, patients will fill in a quality of life questionnaire before they start using the equipment, and then again after 4 weeks and 12 weeks. These brief questionnaires are through simple drop-down menus on the App and take less than 5 minutes to complete.

At the end of 12 weeks, or if individuals leave the study earlier, all the equipment will be returned to the investigating team, to analyse the data.

In addition to the data that we will collect from the digital tools described above, we will also access routine blood tests performed when determined necessary by the liver doctors, as part of the standard of care.

DETAILED DESCRIPTION:
The current Covid Pandemic has necessitated an unusual allocation of healthcare resources which inevitably negatively impacts on resources available to care for patients with chronic diseases including liver disease. This is most marked in those with acute 'decompensation' of cirrhosis, namely the significant subset of patients who develop a rapid decline in liver function and numerous complications including, fluid overload, confusion (encephalopathy), kidney dysfunction and gastrointestinal bleeding.[Jalan et al, J Hepatol 2015; Moreau R et al, Gastroenterology 2013] These patients normally require a regular clinical assessment (every 1-2 weeks) and even when discharged following a recent admission to hospital, have re-admission rates approaching 40% in 8 weeks.[Moranda et al, J Hepatol, 2013] The current unmet need is to institute regular contact with the patient, to avoid further new complications from cirrhosis developing and hospital admission, whilst also avoiding nosocomial (health care setting related) infection with Covid 19 through standard outpatient, scheduled contact. [Tapper EB et al, J Hepatol 2020]

We propose to provide a remote management system for cirrhosis care, which will include remote acquisition of important vital signs such as heart rate, heart rate variability, blood pressure, physical activity and sleep status (through wearable technology), weight, and assessment of higher mental function (smartphone app based tools), all of which are key metrics that are perturbed as cirrhosis decompensation ensues. By efficiently collating this data and linking this to an effective clinical workflow stream based on a platform created for smartphone and clinical user application interfaces, will facilitate improved telemedicine 'consultations' by healthcare providers. This is a novel approach that in this patient cohort, which will allow early detection of signs of complications and rapid triaging of patients who need early direct clinical review, at a time when this is a limited resource. Our solution will help prioritize care whilst limiting risk of COVID-19 infection exposure, and also personalizing this to an individual patient's needs and disease, making this more acceptable and convenient for patients. In the longer term, costs savings will arise through more efficient and streamlined outpatient direct contacts, whilst all patients will receive the priority and regular care input they need.

This is a single centre study at the Royal Free London trust. This is a tertiary liver unit with significant experience in running clinical trials in decompensated cirrhosis. This pilot study has already recruited 20 cirrhosis patients with a known history of decompensation and 20 contemporaneous controls. Potential participants were identified by the PI and/or clinical fellows on the study log, using existing clinic lists and inpatient and discharge lists. The individuals have been monitored using a wrist-watch wearable device, with associated smart weighing scales and blood pressure cuff, along with a smartphone application (including economic smartphone in those patients if not available), to facilitate home monitoring. Currently an interim analysis is being performed on the data collected to assess safety and engagement.

Routine laboratory data was collected in the previous 7 days as part of standard clinical assessment prior to recruitment. Data included liver and kidney function tests and full blood count. The data is logged within the patient historical data on the Cirrhocare App.

All study specific procedures that the participant has undertaken at home were relayed in person during a first study visit meeting, to ensure all the equipment was functional, had been sync'd to work appropriately, and that the participant could operate both the wearables and the Cirrhocare App. The Investigator also provided the participant (and any carer) with written instructions but also a recorded User Guide video on the App. Following patient consent, App set-up, and Cirrhocare Healthkit sync to the patient's (or study provided) phone, and the subsequent patient education steps, the participant, under supervision, performed the baseline App based tests detailed below.

Following the baseline Visit (Visit 1) listed above, the participants were educated with regards to use of their Wearable devices, the use of the Cirrhocare App and the notifications they should expect to receive, such as reminders for the daily measurements required.

Each day, Monday-Friday, between 9am-11am, participants were expected to perform the following measurements:

HRV- as instructed at the baseline visit, and after a brief period of rest when sitting still. This was performed on the Withings move ECG watch after a prompt within the App, which captured their ECG and communicated this to a dedicated Cloud storing daily recordings. The ECG capture was repeated as steps to record 5 minutes of total ECG readings, needed for thorough evaluation of daily HRV. If the participant failed or was unable to complete the task each day after being prompted by the App, they received reminder notifications on their watch and phone to the need for this important data capture. If the participant was unwell and hence felt unable to perform the test, they received a further prompt to enter any symptoms to be communicated to the Investigator team.

BP measurement- participants followed the App prompt to start BP recordings using the supplied Withings cuff. They followed a guide (video clip on the App) that showed placement of the BP cuff on the left arm and when to begin measurement. The recording of BP is automatic through the App and the readings similar to HRV, stored on a Cloud after they are integrated in the App.

Weight measurement - Following the above, the participant was prompted to assess their weight on the supplied Withings scales. They weighed themselves applying bare feet to the scales and with ideally limited loose-fitting clothing so as to standardize daily measurements.

Well-being information: The participants were then prompted to enter their sense of well-being, with drop-down menu prompts (tired, well, unwell, etc.) and the opportunity to input specific symptoms and to request an additional contact.

If the participants had completed the above tasks, they were then next prompted at 8pm to record their daily food and fluid intake through drop-down menus as prompted by the App for simplicity.

The participant was also prompted after the morning measurements, to apply the Stroop Test for encephalopathy as shown to them on visit 1. The App guides them through the completion of the task, which involves naming animals, and then sends the information upon completion of the task to the Cloud.

For all measurements and the Stroop test, the participant received acknowledgement form the App to confirm their data had been logged correctly.

In addition to the tasks requiring direct participant engagement, the Withings Move watch also recorded daily activity as steps, including whether this included vertical climb (stairs) and also sleep patterns (day/night/REM sleep, etc.). This data was collected automatically, which the participant is aware of at the time of consent and helps inform of functional status as well as the development of signs of encephalopathy (i.e increased daytime sleep or inactivity).

Based on daily inputs form participants including measured data as well as food/fluid/sleep and activity data, the physician investigator may have requested a phone call or prompt the participant for further information. For example, if the participant reported new symptoms of a cough or urinary symptoms and has a decrease in HRV or blood pressure, the physician may have prompted the participant to check their temperature with a forehead strip thermometer (also supplied to participants). Another such example might include a check on encephalopathy based on reduced daytime activity or increased sleep or poor Stroop test performance, prompting an additional tele consult.

Physicians also used the outputs that were collated by the App from each participant to gauge the need for additional contact via text messages or phone in addition to the standard scheduled visits, below.

Tele consults were routinely scheduled at week 4, and at week 8 (+/- 5 days), which would historically have been face-to-face appointments pre-COVID 19.

They included assessments of the patient's symptoms, state of encephalopathy (based on conversation and animal naming tests), and assessment of diet and functional status. In addition, routine scheduled blood tests were performed within the week prior to the telephone clinic to inform changes in routine clinical care/treatment. These included, full blood count, liver and kidney function tests, and prothrombin time/INR; C-reactive protein and N-terminal BNP.

Participants also populated their usability questionnaire on the Cirrhocare App at the time of these telephone contacts, and this information was added to any clinician entry on patients' quality of life as discerned by questions during the consultation.

Week 12 involved a face-to-face consultation to assess clinical status by history and clinical examination (i.e. HE, assessment of ascites and oedema, Jaundice, etc) and general symptoms as part of a routine clinical visit for such patients. Patient's HRV, heart rate, BP and weight were re-assessed in the clinic and recorded as the study-end measured variables. Patients were also sent for routine blood test after the appointment and this included; full blood count, liver and kidney function tests, and prothrombin time/INR; C-reactive protein and N-terminal BNP. The results from these routine bloods will be used for assessment of their clinical scores at that time, to reflect their liver decompensation status, namely MELD and EF-CLIF AD scores, as necessary for standard clinical assessment.

During this clinic appointment, a participant Cirrhocare App usability questionnaire was also completed and also a quality-of-life questionnaire.

If the patient requires their routine liver cancer screening ultrasound in the 3-4 month time period when they are participating in the study (done once every 6 months as standard), then this too will be booked routinely. Similarly, most patients undergo routine endoscopic examination for oesophageal varices every year if they have advanced disease. If their screening endoscopy falls within the time frame of their study inclusion, then this too will be booked in routinely. The data from these tests are not specifically required for the study.

As participants are monitored, it is foreseen that some will have events such as increased hepatic encephalopathy (HE), or new infection, as these are expected events in any patient with decompensated cirrhosis. If their monitoring suggests an event may be more likely by for example, changes in activity status (onset of HE) or Increased heart rate and falling blood pressure (potential sepsis), then the Investigator may elect to contact the participant for more information and suggest some advice by an additional telephone call. The outcome of such a contact might trigger a need for further blood tests or even hospital face-to-face assessment, as indicated by the clinical need and individual patient circumstances.

This COVID-19 funded pilot study seeks to evaluate early assessment of usability and feasibility of home monitoring in this advanced cirrhosis population. We are not planning to have further study related visits after 3 months, though patient data on mortality at 3 months and 6 months will be captured for subsequent reporting purposes.

After the last study visit at 12 weeks, patients will return to routine scheduled tele clinic follow-up or face-to-face reviews based on clinical indications (e.g. requirement for ascites drainage), at intervals of around 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age ≥ 18 years old.
2. Cirrhosis defined by standard clinical criteria, ultrasonographic findings and/or histology. Cirrhosis of any aetiology may be included. However, patients with cirrhosis due to autoimmune hepatitis must be on stable corticosteroid dose for ≥3-month period before study inclusion.
3. Child-Pugh A, B patients or Child-Pugh C patients (up to 12 points).
4. Patients with a recent history of cirrhosis decompensation or/and recent discharge from the hospital for an episode of acute cirrhosis decompensation
5. Participants able to give informed consent

Exclusion Criteria:

1. Patients with ACLF according to the criteria published by Moreau et al, Gastro 2013
2. Bacterial infection within 7 days before study inclusion.
3. Gastrointestinal bleeding within 10 days before study inclusion.
4. Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy according to the New-Haven classification. 5. Patients with active hepatocellular carcinoma or history of hepatocellular carcinoma that is in remission for less than six months for uninodular HCC or for less than 12 months for multinodular HCC within Milan criteria.

6. Patients with a history of significant extra hepatic disease with impaired short-term prognosis, including congestive heart failure New York Heart Association Grade III/IV, COPD GOLD >2, chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.

7. Patients with current extra hepatic malignancies including solid tumours and hematologic disorders.

8. Patients with mental incapacity, language barrier, or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.

9.Refusal or inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified by the PI and/or clinical fellows on the study log, using existing clinic lists, and inpatient and discharge lists, containing identifiable personal information, that highlight those patients with decompensated cirrhosis, at risk of further decompensation and who will require regular telephone follow up under the Liver team. The PI and Clinical fellows would normally be reviewing these patients in a routine Out-patient clinic slot - currently by telephone appointments. In addition, patients ready to be discharged from hospital or/and attending day case paracentesis for ascites, will be identified by members of the normal clinical team, to schedule routine follow up.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility and usability of remote monitoring devices | 3 months
  Feasibility and usability of the remote monitoring devices and App will be determined by questionnaires given to the participants at 1, 2 and 3 months of follow-up
Quality of life assessment | 3 months
  A quality of life questionnaire assessed at the outset of the study, will be re-assessed at 1 and 3 months in addition to patient experience reported during direct physician interview.
  This pilot data will be compared to the prior experiences of these patients with telephone follow-up only (or/and hospital visits), during COVID-19.

SECONDARY OUTCOMES:
Complications of cirrhosis | 3 months
  Frequency of well-established complications of cirrhosis in those with previous cirrhosis decompensation will be logged during follow up and include: ascites (fluid overload) and its severity; kidney dysfunction and its severity; hepatic encephalopathy (cognitive dysfunction) and severity; onset of liver related bleeding, and new infections.
Clinical scores of cirrhosis | 3 months
  The clinical scores of cirrhosis decompensation (CLIF-C AD and MELD scores) will be assessed at the trial start and then at 1, 2 and 3 months
Mortality | 6 months
  Mortality at 3 and 6 months will be captured for reporting purposes

CONTACTS AND LOCATIONS:
Overall Officials: Rajeshwar Mookerjee, MBBS, PhD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Jalan R, Pavesi M, Saliba F, Amoros A, Fernandez J, Holland-Fischer P, Sawhney R, Mookerjee R, Caraceni P, Moreau R, Gines P, Durand F, Angeli P, Alessandria C, Laleman W, Trebicka J, Samuel D, Zeuzem S, Gustot T, Gerbes AL, Wendon J, Bernardi M, Arroyo V; CANONIC Study Investigators; EASL-CLIF Consortium. The CLIF Consortium Acute Decompensation score (CLIF-C ADs) for prognosis of hospitalised cirrhotic patients without acute-on-chronic liver failure. J Hepatol. 2015 Apr;62(4):831-40. doi: 10.1016/j.jhep.2014.11.012. Epub 2014 Nov 22. PMID 25463539
- [Background] Morando F, Maresio G, Piano S, Fasolato S, Cavallin M, Romano A, Rosi S, Gola E, Frigo AC, Stanco M, Destro C, Rupolo G, Mantoan D, Gatta A, Angeli P. How to improve care in outpatients with cirrhosis and ascites: a new model of care coordination by consultant hepatologists. J Hepatol. 2013 Aug;59(2):257-64. doi: 10.1016/j.jhep.2013.03.010. Epub 2013 Mar 21. PMID 23523582
- [Background] Tapper EB, Asrani SK. The COVID-19 pandemic will have a long-lasting impact on the quality of cirrhosis care. J Hepatol. 2020 Aug;73(2):441-445. doi: 10.1016/j.jhep.2020.04.005. Epub 2020 Apr 13. PMID 32298769
- [Derived] Gananandan K, Thomas V, Woo WL, Boddu R, Kumar R, Raja M, Balaji A, Kazankov K, Mookerjee RP. Fat mass: a novel digital biomarker for remote monitoring that may indicate risk for malnutrition and new complications in decompensated cirrhosis. BMC Med Inform Decis Mak. 2023 Sep 13;23(1):180. doi: 10.1186/s12911-023-02288-z. PMID 37705043